CLINICAL TRIAL: NCT03543176
Title: Claims-linked Survey Study to Assess Burden of Illness Among Patients Treated With LAMA/LABA vs ICS/LABA Single Inhaler Dual Therapy
Brief Title: Chronic Obstructive Pulmonary Disease (COPD) Dual Therapy Burden of Illness
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: UnitedHealth Group (Industry)
Responsible Party: Sponsor
Other Study IDs: 208782
Record Dates: First submitted 2018-05-18; First posted 2018-06-01 (Actual); Results first posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Cohort; Chronic obstructive pulmonary disease; Observational; GOLD; Claims; Health plan recruitment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — No bio-specimen samples were evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- UMEC/VI: The subjects in this arm had received, UMEC/VI as 62.5/25 microgram (mcg), which is an approved once-daily single inhaler dual LAMA/LABA therapy, given via Ellipta .
  Interventions: Other: UMEC/VI; Other: CAT; Other: mMRC; Device: Ellipta
- FLUT/SAL: The subjects in this arm had received, FLUT/SAL as 250/50 mcg, which is an approved twice-daily single inhaler dual therapy ICS/LABA treatment, given via DISKUS.
  Interventions: Other: FLUT/SAL; Other: CAT; Other: mMRC; Device: Diskus

INTERVENTIONS:
Other: UMEC/VI — UMEC/VI as 62.5/25 mcg, which is a once-daily single inhaler dual therapy, given to subjects, via Ellipta .
  Groups: UMEC/VI
Other: FLUT/SAL — FLUT/SAL as 250/50 mcg, which is a twice-daily single inhaler dual therapy, given to subjects, via Diskus.
  Groups: FLUT/SAL
Other: CAT — Questionnaire used to asses Condition-related well-being, for COPD subjects.
Other: mMRC — Questionnaire used to asses Breathlessness, due to Dyspnea, for COPD subjects.
Device: Ellipta — It is a single once daily, Dry powder Inhaler (DPI), developed for delivery of therapies in COPD subjects.
  Groups: UMEC/VI
Device: Diskus — It is a plastic device containing twice-daily single inhaler dual therapy, developed for delivery of therapies in COPD subjects.
  Groups: FLUT/SAL

SUMMARY:
The main purpose of the study is to assess the burden of illness for, COPD using both patient-reported symptom burden and claims-based economic burden, among the subjects treated with single-inhaler dual therapy treatments, Fluticasone/Salmeterol FLUT/SAL; Advair) or Umeclidinium/Vilanterol (UMEC/VI; Anoro) to support Global Initiative for Chronic Lung Disease (GOLD) category B recommendations. The study will use a health plan recruitment strategy and subject's will be recruited using Optum's health plan recruitment strategy to collect information relating to the subject's condition history, current treatment, smoking history, symptoms and symptom severity (Modified Medical Research Council Dyspnoea Scale [mMRC] and COPD Assessment Test [CAT]), and demographic and sociodemographic characteristics. A total of 2700 subject's, are planned to be enrolled in the study to reach the target evaluable sample size, n=770 subjects. Following completion of data collection, results of the survey, will be merged with claims data, covering the 12-month Baseline period for analysis. Pharmacy and medical claims data, will be used to calculate all-cause and COPD-related health care utilization and costs, treatment patterns, and Baseline clinical characteristics. The study duration is estimated to be of 12-months.

ELIGIBILITY:
Inclusion Criteria:

* >=2 International Statistical Classification of Diseases and Related Health Problems (ICD)-10-CM diagnosis codes for COPD at least 30 days apart during the 12 month period prior to sample identification.
* Diagnosis codes J40-J44 will be included.
* >=1 pharmacy claim for UMEC/VI or FLUT/SAL single-inhaler dual therapy during Baseline.
* Age >= 65 years.
* Self-reported health care provider diagnosis of COPD.
* Self-reported prescription for FLUT/SAL or UMEC/VI.
* 12 months of continuous enrollment during the Baseline period.
* Ability to complete the study survey in English.

Exclusion Criteria:

* >=2 ICD-10-CM diagnosis codes for asthma at least 30 days apart during the, 12 month period, prior to sample identification.
* Claims for both UMEC/VI and FLUT/SAL in the 6 months, closest to sample identification.
* Claims for triple therapy (Inhaled Corticosteroid [ICS] + Long-acting Antimuscarinic [LAMA] + Long-acting Beta-agonist [LABA] during the Baseline period.
* Evidence of lung cancer diagnosis and/or treatment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study will include Medicare Advantage (Medicare) health plan members with evidence of COPD, in the 12 months prior to sample identification and evidence of treatment with UMEC/VI or FLUT/SAL, single-inhaler dual therapy in the six months prior to sample identification. All adults (male and female) subjects with age, greater than or equal to 65 years will be included.
Sampling Method: Non-Probability Sample
Enrollment: 789 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2019-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Date Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available, within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided, after a research proposal is submitted and has submitted approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided, for an initial period of 12 months but an extension can be granted, when justified for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This cross-sectional observational survey study aimed to assess symptom burden and Baseline clinical and economic characteristics in chronic obstructive pulmonary disease (COPD) participants treated with single-inhaler dual therapies in adult Medicare Advantage (MA) enrollees with COPD diagnosis and treatment.
Pre-assignment Details: A total of 789 claims linked analytic participants were enrolled in the study.
Groups:
- Umeclidinium/Vilanterol: Participants in this arm received Umeclidinium/Vilanterol as 62.5/25 microgram (mcg), which is an approved once-daily single inhaler dual Long-acting anti-muscarinic (LAMA)/ Long-acting beta-agonist (LABA) therapy, given via Ellipta
- Fluticasone /Salmeterol: Participants in this arm received Fluticasone/Salmeterol as 250/50 mcg, which is an approved twice-daily single inhaler dual therapy Inhaled Corticosteroid (ICS)/LABA treatment, given via DISKUS.
Period: Overall Study
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Started | 392 | 397
Completed | 392 | 397
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol | Total
Number analyzed (Participants) | 392 | 397 | 789
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.69 (6.01) | 75.52 (6.10) | 75.60 (6.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 222 | 423
  Male | 191 | 175 | 366
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-minority | 357 | 351 | 708
  Black/Asian/Other Race, Minority | 35 | 44 | 79
  Missing | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Reported COPD Symptom Burden- Measured Using COPD Assessment Test (CAT) Questionnaire
Description: The CAT questionnaire is an 8-item questionnaire on a 0-5 point scale with higher values indicating greater impact of COPD. The item response values of CAT are summed to produce a single score that ranges from 0-9 (low impact), 10-20 (medium impact), 21-30 (high impact) and 31-40 (very high impact). Respondents were allowed to have up to two missing CAT items. If one or two items were missing, the total score was set to the average of the non-missing item scores. Percentage of participants reporting low, medium, high and very high impact COPD symptom burden on CAT scale has been presented. All enrolled Population comprises of all participants with claims >= 1.
Time Frame: Day 1
Population: All enrolled Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Percentage of participants
  Low impact (0-9) | 13.27 | 11.34
  Medium impact (10-20) | 51.28 | 43.58
  High impact (21-30) | 30.36 | 35.01
  Very high impact, (31-40) | 5.10 | 10.08
Statistical Analysis 1: Comparison: Umeclidinium/Vilanterol vs Fluticasone /Salmeterol; Test type: Other; p = 0.448, Fisher Exact — P-value for low impact of COPD is presented
Statistical Analysis 2: Comparison: Umeclidinium/Vilanterol vs Fluticasone /Salmeterol; Test type: Other; p = 0.033, Fisher Exact — P-value for medium impact of COPD is presented
Statistical Analysis 3: Comparison: Umeclidinium/Vilanterol vs Fluticasone /Salmeterol; Test type: Other; p = 0.172, Fisher Exact — P-value for high impact of COPD is presented
Statistical Analysis 4: Comparison: Umeclidinium/Vilanterol vs Fluticasone /Salmeterol; Test type: Other; p = 0.010, Fisher Exact — P-value for very high impact of COPD is presented

2. Primary Outcome: Percentage of Participants That Reported COPD Symptom Burden- Measured Using Modified Medical Research Council (mMRC) Dyspnea Scale
Description: Breathlessness was assessed using the mMRC, a single item (0-4) scale assessing current level of dyspnea. The mMRC comprised of five statements that describe almost the entire range of respiratory disability from none (Grade 0) to almost complete incapacity (Grade 4). The score (Grade) was the number that best fit the participant's level of activity. The mMRC categorized participants into low dyspnea (Grades 0-1) and high dyspnea (Grades 2-4).
Time Frame: Day 1
Population: All enrolled Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Percentage of participants
  Grades (0-1) | 51.79 | 46.85
  Grades (2-4) | 48.21 | 53.15
Statistical Analysis 1: Comparison: Umeclidinium/Vilanterol vs Fluticasone /Salmeterol; Test type: Other; p = 0.176, Fisher Exact — P-value for breathlessness reported in COPD assessed using mMRC is presented

3. Secondary Outcome: Mean Baseline Comorbidity Burden Score Using Quan-Charlson-clinical Characteristics
Description: A comorbidity score was calculated based on the presence of diagnosis codes on medical claims in the Baseline period. The mean score has been presented. the scores was categorized into the following groups: one to two, three to four and five or more.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Scores on a scale | 2.53 (1.91) | 2.49 (1.74)
Statistical Analysis 1: Comparison: Umeclidinium/Vilanterol vs Fluticasone /Salmeterol; Test type: Other; p = 0.732, t-test, 2 sided — P-value for Baseline comorbidity burden score was calculated

4. Secondary Outcome: Mean Count of Unique Medications-Baseline All Cause Utilization
Description: A count of unique medications filled in the 12-month Baseline period was calculated. The mean values has been presented.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Mean (Standard Deviation); unit: Medications
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Medications | 13.39 (5.99) | 14.52 (6.67)
Statistical Analysis 1: Comparison: Umeclidinium/Vilanterol vs Fluticasone /Salmeterol; Test type: Other; p = 0.013, t-test, 2 sided — P-value for count of unique medications was calculated

5. Secondary Outcome: Mean Total Number of Medications Dispensing-Baseline All Cause Utilization
Description: A count of unique dispensing's for all medications filled in the 12-month Baseline period was calculated.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Mean (Standard Deviation); unit: Medications dispensing
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Medications dispensing | 43.55 (26.15) | 46.22 (29.46)
Statistical Analysis 1: Comparison: Umeclidinium/Vilanterol vs Fluticasone /Salmeterol; Test type: Other; p = 0.178, t-test, 2 sided — P-value for total number of medications dispensing was calculated

6. Secondary Outcome: Percentage of Participants With All Cause Healthcare Resource Utilization
Description: Binary indicators and counts of ambulatory (physician office and hospital outpatient) visits, emergency department (ED) visits, and inpatient stays were calculated in the 12-month Baseline period. Percentage of participants with inpatient stays, emergency room visits, ambulatory visits, office visits and outpatient visits in Baseline period has been presented.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Percentage of participants
  Inpatient stays | 28.83 | 31.49
  Emergency room visits | 44.64 | 50.38
  Ambulatory visits | 100.00 | 100.00
  Office visits | 98.72 | 97.98
  Outpatient visits | 84.69 | 87.41

7. Secondary Outcome: Mean Number of Inpatient Admissions -Baseline All Cause Utilization Counts
Description: Mean number of inpatient admissions during the 12 months Baseline period has been presented.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Mean (Standard Deviation); unit: Inpatient Hospital Admissions
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Inpatient Hospital Admissions | 0.40 (0.76) | 0.47 (0.85)

8. Secondary Outcome: Length of Stay in Hospital-Baseline All Cause Utilization Counts
Description: Binary indicators and counts of inpatient stays were calculated in the 12-month Baseline period. Length of stay during the 12 months Baseline period has been presented.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Days | 3.51 (10.09) | 3.95 (9.57)

9. Secondary Outcome: Mean Number of Emergency Room, Ambulatory, Office and Outpatient Visits-Baseline All Cause Utilization Counts
Description: Binary indicators and counts of ambulatory (physician office and hospital outpatient) visits and ED visits were calculated in the 12-month Baseline period. Mean number of emergency room, ambulatory, office and outpatient visits during the 12 months Baseline period has been presented.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Mean (Standard Deviation); unit: Hospital visits
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Hospital visits
  Emergency room visits | 0.91 (1.53) | 1.18 (1.90)
  Ambulatory visits | 26.79 (18.10) | 25.51 (17.76)
  Office visits | 16.70 (12.34) | 15.54 (12.42)
  Outpatient visits | 10.12 (11.45) | 10.04 (10.34)

10. Secondary Outcome: Mean Total Baseline All Cause Healthcare Costs
Description: Consumer Price Index-adjusted costs were assessed for the 12-month Baseline period. Costs were calculated as total costs, pharmacy costs, and medical costs; medical costs include ambulatory (physician office and hospital outpatient) costs, emergency costs, inpatient costs, and other costs. Mean total all cause healthcare costs that includes medical costs and pharmacy costs during the 12 months Baseline period has been presented.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
US Dollars | 19915.66 (31213.46) | 17591.88 (21533.79)

11. Secondary Outcome: Mean Count of Unique COPD Medications-Baseline COPD Medication
Description: A count of unique COPD medications filled in the 12-month Baseline period was calculated. The mean values have been presented.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Mean (Standard Deviation); unit: Medications
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Medications | 0.99 (0.10) | 0.99 (0.09)
Statistical Analysis 1: Comparison: Umeclidinium/Vilanterol vs Fluticasone /Salmeterol; Test type: Other; p = 0.692, t-test, 2 sided — P-value for count of unique COPD medications was calculated

12. Secondary Outcome: Mean Total Number of COPD Medications Dispensing-Baseline COPD Medications
Description: A count of unique COPD dispensings for all medications filled in the 12-month Baseline period was calculated.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Mean (Standard Deviation); unit: Medications dispensing
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Medications dispensing | 2.50 (1.40) | 1.76 (1.11)
Statistical Analysis 1: Comparison: Umeclidinium/Vilanterol vs Fluticasone /Salmeterol; Test type: Other; p < 0.001, t-test, 2 sided — P-value for total number of COPD medications dispensing was calculated

13. Secondary Outcome: Percentage of Participants With COPD Related Baseline Healthcare Resource Utilization
Description: Binary indicators and counts of ambulatory (physician office and hospital outpatient) visits, ED visits, and inpatient stays were calculated in the 12-month Baseline period. Utilization defined was considered COPD-related when a diagnosis code for COPD is in the primary position. Percentage of participants with inpatient stay, emergency room, ambulatory, office and outpatient visits during the 12-months Baseline period has been presented.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Percentage of participants
  Inpatient stay | 13.78 | 13.60
  Emergency room visits | 10.71 | 16.37
  Ambulatory visits | 83.93 | 75.57
  Office visits | 77.30 | 61.46
  Outpatient visits | 39.03 | 28.97

14. Secondary Outcome: Mean Number of Inpatient Admissions -Baseline COPD Related Utilization Counts
Description: Mean number of Baseline COPD related inpatient admissions during the 12 months Baseline period has been presented.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Mean (Standard Deviation); unit: Admissions
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Admissions | 0.17 (0.50) | 0.17 (0.48)

15. Secondary Outcome: Length of Inpatient Stay-Baseline COPD Related Utilization Counts
Description: Binary indicators and counts of inpatient stays were calculated in the 12-month Baseline period. Baseline COPD related length of inpatient stay during the 12 months Baseline period has been presented.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Days | 2.02 (8.34) | 1.57 (6.18)

16. Secondary Outcome: Mean Number of Emergency Room, Ambulatory, Office and Outpatient Visits-Baseline COPD Related Utilization Counts
Description: Binary indicators and counts of ambulatory (physician office and hospital outpatient) visits and ED visits were calculated in the 12-month Baseline period. Mean number of Baseline COPD related emergency room, ambulatory, office and outpatient visits during the 12 months Baseline period has been presented.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Mean (Standard Deviation); unit: Hospital visits
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Hospital visits
  Emergency room visits | 0.16 (0.55) | 0.21 (0.54)
  Ambulatory visits | 3.21 (2.88) | 2.38 (3.02)
  Office visits | 2.18 (2.21) | 1.47 (1.72)
  Outpatient visits | 1.03 (1.78) | 0.91 (2.25)

17. Secondary Outcome: Mean Total Baseline COPD-related Healthcare Costs
Description: Consumer Price Index-adjusted costs were assessed for the 12-month Baseline period. Costs was calculated as total costs, pharmacy costs, and medical costs; medical costs include ambulatory (physician office and hospital outpatient) costs, emergency costs, inpatient costs, and other costs. Costs defined was considered COPD-related if the claim has a diagnosis code for COPD in the primary position or is for a medication used to treat COPD. Mean total Baseline COPD related healthcare costs that includes medical costs and pharmacy costs during the 12 months Baseline period has been presented.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
US Dollars | 5008.86 (11551.58) | 3797.44 (7246.79)

18. Secondary Outcome: Number of Participants With Atleast One Baseline COPD Exacerbation
Description: Whether the participant has evidence of a COPD exacerbation during the 12-month Baseline period was captured. A moderate COPD exacerbation was defined as either an emergency room visit with the primary diagnosis of COPD and/or an ambulatory visit with the primary diagnosis of COPD. The COPD-related qualifying emergency room or ambulatory event must also have a dispensing of antibiotics or systemic corticosteroids +/- 5 days from the date of service of the emergency room or ambulatory event. A severe COPD exacerbation was defined as a hospitalization with a primary diagnosis code of COPD. The count of participants with atleast one COPD exacerbation has been presented.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Participants | 164 | 184

19. Secondary Outcome: Percentage of Participants in Each Global Initiative for Chronic Lung Disease (GOLD) Category Classification
Description: The GOLD categories were classified based on CAT and mMRC scores. GOLD A includes participants reporting COPD CAT symptoms score <10 and mMRC as 0-1; GOLD B includes participants reporting CAT symptom score >=10 and mMRC as >=2; GOLD C includes participants reporting exacerbation history as >=2 or >=1 leading to hospitalization; GOLD D includes participants reporting exacerbation history as 0 or 1 and not leading to hospitalization. The number of participants in each GOLD category of symptom burden and exacerbation, was presented. The calculation used was count of COPD exacerbations during the Baseline combined with CAT total score and mMRC score to create mutually exclusive counts for each category.
Time Frame: 12 months
Population: All enrolled Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
Number analyzed (Participants) | 392 | 397
Percentage of participants
  GOLD A with mMRC only | 43.37 | 37.28
  GOLD B with mMRC only | 33.42 | 38.54
  GOLD C with mMRC only | 8.42 | 9.57
  GOLD D with mMRC only | 14.80 | 14.61
  GOLD A with CAT only | 11.73 | 9.82
  GOLD B with CAT only | 65.05 | 65.99
  GOLD C with CAT only | 1.53 | 1.51
  GOLD D with CAT only | 21.68 | 22.67
  GOLD A with mMRC and CAT | 10.20 | 9.82
  GOLD B with mMRC or CAT | 66.58 | 65.99
  GOLD C with mMRC and CAT | 1.02 | 1.51
  GOLD D with mMRC or CAT | 22.19 | 22.67

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were not collected as this is a cross-sectional retrospective claims study that utilized enrollment, medical, and pharmacy records from Optum's proprietary research claims database (ORD) without a GlaxoSmithKline drug of interest.
Description: AEs and serious adverse events (SAEs) were not collected.
Arm/Group | Umeclidinium/Vilanterol | Fluticasone /Salmeterol
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT03543176/Prot_SAP_000.pdf